CLINICAL TRIAL: NCT04949035
Title: Assessment of Mental Status and Quality of Life of Patients Admitted to the Rehabilitation Unit After COVID-19 Hospitalization
Brief Title: Mental Status and Quality of Life of Post-COVID-19 Patients
Status: Completed | Type: Observational
Sponsor: The Opole University of Technology (Other)
Responsible Party: Principal Investigator, Sebastian Rutkowski, Assistant Professor, The Opole University of Technology
Other Study IDs: COVID-19 Pre-
Record Dates: First submitted 2021-07-01; First posted 2021-07-02 (Actual); Last update posted 2021-08-09 (Actual); Status verified 2021-08

CONDITIONS: Covid19
Keywords: quality of life; HADS; rehabilitation; anxiety
MeSH Terms: conditions — COVID-19; Anxiety Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- COVID-19 survivors
  Interventions: Diagnostic Test: Assessment of mental state and quality of life

INTERVENTIONS:
Diagnostic Test: Assessment of mental state and quality of life — Patients qualified for rehabilitation will be assessed for stress levels as well as symptoms of anxiety and depression and quality of life before rehabilitation began

SUMMARY:
The current SARS-CoV-2 virus pandemic has already affected the lives of every person on earth. Most of the information given in the media on a daily basis focuses on the pandemic aspects. Fear of getting sick arises in the population, and once infection occurs, numerous concerns arise over the course of the disease. For some patients, hospitalization and subsequent rehabilitation is needed due to complications from the disease. Besides the aspect of treating patients physically from the disease, the psychological aspects that often accompany patients during and after the disease are not addressed. Depressive and anxiety symptoms can follow patients for many years and can affect their quality of life. Thus, the purpose of this project is to assess the mental status of patients prior to the inpatient rehabilitation program

DETAILED DESCRIPTION:
Patients with COVID-19 or post-COVID-19 will have a need for rehabilitation during and directly after hospitalization. Data on safety and efficacy are lacking, as the number of COVID-19 survivors has increased rapidly. The Convergence of Opinion on Recommendations and Evidence process was used to make interim recommendations for the in-hospital rehabilitation and post-hospital phase in patients with COVID-19 and post-COVID-19 patients, respectively. The International Task Force (ITS) was established, including the European Respiratory Society (ERS) and key opinion leaders from the American Thoracic Society (ATS), as well as key opinion leaders in the field of lung rehabilitation. In its report, the ITS identified recommendations for the rehabilitation of patients with COVID-19 and post-COVID-19 patients. Majority of the experts recommended strongly (71%) or conditionally (24%) for COVID-19 survivors with symptoms of psychological distress at 6-8 weeks after discharge from the hospital receiving a formal psychological assessment. Therefore, this project aims to evaluate the mental status and quality of life of patients admitted to the rehabilitation unit, after COVID-19 hospitalization.

In our project, we intend to answer the following questions:

* What is the severity of depressive symptoms in individuals who have suffered COVID-19 ?
* What is the severity of anxiety symptoms in individuals who have suffered COVID-19 ?
* What is the level of perceived stress in individuals who have suffered COVID-19 ?
* What is the quality of life of people in individuals who have suffered COVID-19 ?

ELIGIBILITY:
Inclusion Criteria:

* Previously hospitalized for SARS-CoV-2 infection;
* Pulmonary rehabilitation conducted in ward settings

Exclusion Criteria:

* Inability to self-complete the research questionnaires;
* Presence of the following issues at the time of the examination or in the medical data: disturbances of consciousness, psychotic symptoms or other serious psychiatric disorders
* Initiation of psychiatric treatment during the research project;
* Patient's refusal at any stage of the research project.

Ages: 30 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: COVID-19 caused by SARS-CoV-2 has led to a global public health crisis. Clinical symptoms of patients with COVID-19 infection include fever, sore throat, coughing, fatigue, or gastrointestinal infections, which can appear in a smaller population of patients. In more severe cases, respiratory failure symptoms, as well as heart and kidney damage, may occur. This can happen especially in the elderly and in people with other concomitant chronic diseases. Furthermore, the COVID-19 pandemic gives rise to new psychosocial and emotional stressors for recovering patients, including social isolation, physical distancing, loss of employment and uncertainties about the future. Remarkably, many mental problems will continue long after the pandemic is over, some of which will only begin to emerge in the near future.
Sampling Method: Non-Probability Sample
Enrollment: 147 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-05-28 (Actual); Study Completion 2021-06-07 (Actual)

PRIMARY OUTCOMES:
Hospital Anxiety and Depression Scale (HADS) | 15 minutes
  The Hospital Anxiety and Depression Scale (HADS) is a fourteen-item scale scoring from 0 to 3 for each item. The first seven items relate to anxiety (HADS-A), and the remaining seven items relate to depression (HADS-D). The global scoring ranges from 0 to 42 with a cut-off point of 8/21 for anxiety and 8/21 for depression. The higher the score, the greater anxiety or depression symptoms. HADS will be performed at the beginning and after four weeks of treatment.
Perceived stress scale (PSS-10) | 15 minutes
  The Perceived Stress Scale (PSS) is the most widely used psychological instrument for measuring the perception of stress. It is a measure of the degree to which situations in one's life are appraised as stressful. Items were designed to tap how unpredictable, uncontrollable, and overloaded respondents find their lives.
WHOQOL-BREF | 10 minutes
  The WHOQOL-BREF is a shorter version of the WHOQOL-100. Both were developed by the World Health Organisation (WHO) and published in 1995. It was developed over several years and from 15 centres around the world. The questions stem from multiple statements about quality of life, health and well-being from people with and without disease, and health professionals. It has been tested for reliability and validity. The WHOQOL-BREF is a self-administered questionnaire comprising 26 questions on the individual's perceptions of their health and well-being over the previous two weeks. Responses to questions are on a 1-5 Likert scale where 1 represents "disagree" or "not at all" and 5 represents "completely agree" or "extremely".

SECONDARY OUTCOMES:
Six-Minute Walk Test (6MWT) | 10 minutes
  The six-minute walk test measures the distance a patient is able to walk over a total of six minutes on a firm, flat surface. The aim is for the patient to walk as far as possible in six minutes. The patient is allowed to self-pace and rest as needed as they traverse back and forth along a marked walkway.
Spirometry Test | 20 minutes
  The patient is asked to take the deepest breath they can, and then exhale into the sensor as hard as possible, for as long as possible, preferably at least 6 seconds. It is sometimes directly followed by a rapid inhalation, in particular when assessing possible upper airway obstruction.

CONTACTS AND LOCATIONS:
Overall Officials: Joanna Szczepańska-Gieracha, Prof, Study Director — University School of Physical Education, Department of Physiotherapy, Wroclaw, Poland; Sebastian Rutkowski, PhD, Study Chair — The Opole University of Technology, Opole, Poland; Patryk Szary, MSc, Principal Investigator — University School of Physical Education, Department of Physiotherapy, Wroclaw, Poland
Locations (1):
- The Ministry of the Interior and Administration Hospital, Głuchołazy, Poland

IPD SHARING:
Plan to Share IPD: No